CLINICAL TRIAL: NCT06488664
Title: Multicenter International Single-blind Randomized Comparative Clinical Study of the Efficacy and Safety of GNR-068 (45 mg) and Stelara® (45 mg) and Assessment of the Safety, Tolerability and Long-term Effectiveness of GNR-068 in Patients With Moderate and Severe Forms of Plaque Psoriasis
Brief Title: An Efficacy and Safety Study of GNR-068 (Ustekinumab Biosimilar) and Stelara® in the Treatment of Patients With Moderate to Severe Plaque Psoriasis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKM-PS-III
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Plaque Psoriasis
Keywords: ustekinumab; humanized monoclonal antibodies; safety; plaque psoriasis; equivalence; biosimilar; PASI (Psoriasis Area and Severity Index); BSA (Body Surface Area); DLQI (Dermatological Life Quality Index); PGA (Physician's Global Assessment); immunogenicity
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GNR-068 (JSC "GENERIUM", Russia) (Experimental): Test drug
  Interventions: Biological: GNR-068
- Stelara® (manufacturer Silag AG, Switzerland) (Active Comparator): reference drug
  Interventions: Biological: Stelara®

INTERVENTIONS:
Biological: GNR-068 — GNR-068 was administered subcutaneously at weeks 0 and 4 weeks then every 12 weeks thereafter until week 52.
  Other Names: ustekinumab biosimilar
  Arms: GNR-068 (JSC "GENERIUM", Russia)
Biological: Stelara® — Stelara® was administered subcutaneously at weeks 0 and 4 weeks then every 12 weeks thereafter until week 28 and then all patients receive GNR-068 45 mg until week 52.
  Other Names: ustekinumab
  Arms: Stelara® (manufacturer Silag AG, Switzerland)

SUMMARY:
This is a randomized single-blind comparative parallel group efficacy and safety study of ustekinumab biosimilar GNR-068 (45 mg) and reference product Stelara® (45 mg) in the treatment of patients with moderate and severe forms of plaque psoriasis. Participants received a subcutaneous dose of ustekinumab 45 mg (GNR-068 or Stelara®) at weeks 0 and 4 weeks then every 12 weeks thereafter until week 28 and then all patients receive GNR-068 45 mg. For patients with partially respond to the initial regimen the regimen can be adjusted.

DETAILED DESCRIPTION:
The drug GNR-068 (INN: ustekinumab) is being developed as a biosimilar to the drug Stelara®, solution for subcutaneous administration (Silag AG, Switzerland).

Preclinical studies and early phase clinical studies suggest that interleukins-12 (IL-12) and -23 (IL-23), two molecules that are part of the communication network in the immune system, may play an important role in psoriasis. Ustekinumab is a monoclonal antibody directed against IL-12 and IL-23. This is a randomized, single blind, parallel-group, multicenter study to determine the effectiveness and safety of ustekinumab biosimilar GNR-068 administered subcutaneously as compared with Stelara® in patients with moderate to severe plaque-type psoriasis. Patients receive GNR-068 45 mg or Stelara 45 mg administered subcutaneously at weeks 0 and 4 weeks then every 12 weeks thereafter until week 28, thereafter until week 52 all patients receive GNR-068. For patients who partially respond to the initial regimen, the dose can be adjusted to 90 mg and then the interval can be adjusted to every 8 weeks. The study included a screening period, comparative treatment period, non-comparative treatment period, follow up period. Allocation of patients to treatment groups was carried out by randomization in a ratio of 1:1. 422 patients (211 to each study groups) were randomized.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in the study.
* Men and women 18-75 years of age, inclusive, at the time of signing the informed consent form.
* Patients diagnosed with plaque psoriasis at least 6 months before screening:

  1. Moderate or severe form of the disease, which is defined as: PASI index ≥12, body surface area (BSA) affected by plaque psoriasis, ≥10%, PGA scale score ≥3 (on a scale from 0 to 4).
  2. Presence of indications for systemic therapy, defined as inadequate control of the disease against the background of: local treatment (including local glucocorticosteroids) and/or phototherapy and/or lack of clinical effect from the use of other systemic methods.
  3. It is acceptable to carry out basic therapy for psoriatic arthritis at a stable dose for ≥ 4 weeks before screening: prednisolone at a dose of ≤10 mg per day, NSAIDs, methotrexate at a dose of ≤15 mg per week, sulfasalazine at a dose of 2.0 g per day.
* Body weight less than 100 kg.
* If it is necessary to take drugs that worsen the course of psoriasis (beta blockers, calcium channel blockers, lithium drugs, etc.): a stable dose of these drugs for ≥ 4 weeks before randomization.
* Consent of women of childbearing age, women in menopause lasting less than 2 years and male patients to comply with adequate methods of contraception throughout the study and for 3 months after the end of ustekinumab therapy.
* Patients should not be donors of blood or its components 30 days before inclusion in the study and not become donors of blood or its components throughout the study and for 3 months after its completion.

Exclusion Criteria:

* Types of psoriasis other than plaque, except for concomitant psoriatic arthritis.
* History of therapy with ustekinumab or any therapy aimed at IL-12 or IL-23 (briakinumab, guselkumab, tildrakizumab).
* Therapy with TNF-alpha inhibitors or any other genetically engineered biological drugs within 3 months before randomization.
* Conducting other systemic therapies (including cyclosporine, acitretin, methotrexate, UV and PUVA therapy) within 1 month before randomization.
* Treatment with leflunomide for 6 months before randomization.
* Spread of the inflammatory process involving the gastrointestinal tract (inflammatory bowel diseases), the organ of vision (uveitis, iridocyclitis), musculoskeletal structures (high activity of psoriatic arthritis, osteoarthritis, uncontrolled against the background of basic therapy (clause 3 Inclusion criteria) ).
* Major surgery (including joint surgery) within 8 weeks before the start of the study or elective surgery within 6 months after the start of the study.
* A history of an adverse drug reaction to any of the components of the study drug or a reference drug.
* Immunization with any live or live attenuated vaccine within 1 month before the first dose of the study drug or comparator drug.
* A history of a disease associated with the accumulation of immune complexes that may distort the assessment of the effectiveness of ustekinumab therapy (including serum sickness, systemic lupus erythematosus, rheumatoid arthritis, polymyositis, scleroderma, Sjogren's syndrome, vasculitis, cryoglobulinemia).
* Concomitant diseases and conditions that, in the opinion of the Investigator and/or Sponsor, jeopardize the safety of the patient during participation in the study, or which will influence the analysis of safety data.
* Active systemic infection (bacterial, viral or fungal) within 14 days before signing the informed consent.
* Pregnancy or breastfeeding.
* History of tuberculosis, positive/doubtful result of screening for tuberculosis infection (tuberculosis allergen test or IGRA test or fluorography results). Inclusion of such patients is possible if effective specific treatment for tuberculosis infection has been carried out and there is a conclusion from a phthisiatrician about the possibility of ustekinumab therapy.
* Participation in clinical trials of drugs less than 5 half-lives of the study drug before signing the informed consent.
* Positive test for hepatitis B or C, HIV or syphilis.
* Unwillingness or inability to comply with the recommendations prescribed by this protocol.
* Identification during screening of other diseases/conditions not listed above that, in the opinion of the physician-researcher, prevent the inclusion of the patient in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with Psoriasis Area and Severity Index (PASI) Score of 75 Percent or Above | Week 12
  PASI is a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score. The scale ranges from 0 (best) to 72 (worst).

SECONDARY OUTCOMES:
The proportion of patients achieving PASI50/75/90/100 | Week 60
  PASI is a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
Time to reach PASI50, PASI75, PASI90, PASI100 | Week 60
  PASI is a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
Area under the curve (AUC) of PASI | Week 60
  PASI is a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
The proportion of partial responders (ie, patients achieving ≥50% but <75% improvement in PASI compared to baseline) | Week 60
  PASI is a widely used tool for the measurement of severity of psoriasis. This is a test of how bad a person's psoriasis is. The scale combines redness, scaling, and thickness, as well as overall body involvement to determine the PASI score. The scale ranges from 0 (best) to 72 (worst).
Changes in the BSA index | Week 60
  Using the BSA (Body Surface Area) index, the surface area of the skin affected by psoriasis is assessed. BSA is measured in %. To determine the area of psoriatic skin lesions the "palm" rule is applicable. On the scalp, the affected area the size of one palm is assumed to be 10%, the torso - 3.3%, the upper extremities - 5%, the lower extremities - 2.5% of the area of the anatomical region of the body. To calculate the total BSA, each reported percentage must be multiplied by the corresponding factor of the corresponding body region (head = 0.1, torso = 0.3, upper extremities = 0.2, lower extremities = 0.4). The resulting four percentage values (percentage of skin affected by psoriasis on the scalp, upper extremities, trunk, and lower extremities) will be summed to estimate the BSA index.
Changes in PGA | Week 60
  The PGA is 7-point scale used in clinical trials of various diseases. In this the physician checks the state of the disease and gives them score from 0 (clear) to 5 (severe).
Changes in the intensity of itching on the visual analogue scale (VAS) | Week 60
  The intensity of itching is carried out at all visits using a visual analogue scale (VAS), where the left end of the line is 0 = no itching, the right end of the line is 10 = intense itching
Changes in quality of life, assessed using the Dermatology Life Quality Index (DLQI) | Week 60
  The DLQI is a 10-item questionnaire, that in addition to evaluating overall quality of life, can be used to assess 6 different aspects that may affect quality of life: symptoms and feelings, daily activities, leisure, work or school performance, personal relationships, and treatment. Scores range from 0 (no impairment in quality of life) to 30 (most impairment in quality of life).
The proportion of patients who dropped out of the study due to lack of sufficient therapeutic response | Week 60
  Treatment failure is assessed as no effect within 28 weeks (PASI response <50%)

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — JSC GENERIUM
Locations (34):
- Russia (34):
  - Federal State Budgetary Educational Institution of Higher Education "Altai State Medical University" of the Ministry of Health of the Russian Federation, Barnaul, Barnaul
  - State budgetary healthcare institution "Chelyabinsk Regional Clinical Dermatovenerological Dispensary", Chelyabinsk, Chelyabinsk Oblast
  - Limited Liability Company "Ecology of Health", Chelyabinsk, Chelyabinsk Oblast
  - State budgetary institution of the Sverdlovsk region "Ural Research Institute of Dermatovenereology and Immunopathology", Yekaterinburg, Ekaterinburg
  - Limited Liability Company "Alliance Biomedical - Ural Group", Izhevsk, Izhevsk
  - Federal State Budgetary Educational Institution of Higher Education "Kirov State Medical University" of the Ministry of Health of the Russian Federation (FSBEI HE Kirov State Medical University of the Ministry of Health of Russia)), Kirov, Kirov Oblast
  - Limited Liability Company "Available Polyclinic", Murino, Leningradskaya Oblast'
  - State health care institution "Regional Dermatovenerological Dispensary", Lipetsk, Lipetsk Oblast
  - Limited Liability Company "OLLA-MED", Moscow, Moscow
  - Federal State Budgetary Institution "Research Institute of Rheumatology named after V.A. Nasonova", Moscow, Moscow
  - Limited Liability Company "Firma ORIS", Moscow, Moscow
  - State budgetary healthcare institution of the city of Moscow "Moscow Scientific and Practical Center of Dermatovenereology and Cosmetology of the Moscow Health Department", Moscow, Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Russian University of Medicine" of the Ministry of Health of the Russian Federation (FSBEI HE "Russian University of Medicine" of the Ministry of Health of Russia), Moscow, Moscow
  - State budgetary healthcare institution of the Moscow region "Moscow Regional Research Clinical Institute named after M.F. Vladimirsky", Moscow, Moscow
  - Limited Liability Company "Family Clinic No. 4", Korolyov, Moscow Oblast
  - Limited Liability Company "Medical Center "Healthy Family", Novosibirsk, Novosibirsk Oblast
  - Federal State Budgetary Educational Institution of Higher Education Orenburg State Medical University of the Ministry of Health of Russia, Orenburg, Orenburg Oblast
  - State budgetary institution of the Ryazan region "Regional clinical dermatovenerological dispensary", Ryazan, Ryazan Oblast
  - Limited Liability Company "Clinic of Skin Diseases Pierre Wolkenstein", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "International Medical Center", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Medical Technologies" LLC "Medical Technologies", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Health Energy", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Interleukin", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Institute of Medical Research", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "PiterKlinika", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "ArsVite North-West", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Curator", Saint Petersburg, Sankt-Peterburg
  - Private medical institution "Euromedservice", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "MEDINET", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "SB Clinic of Cosmetology", Saratov, Saratov Oblast
  - Regional state budgetary healthcare institution "Smolensk Dermatovenerological Dispensary", Smolensk, Smolensk Oblast
  - Limited Liability Company Medical Center "Azbuka Health", Kazan', Tatarstan Republic
  - State Budgetary Healthcare Institution Ulyanovsk area Clinical Hospital, Ulyanovsk, Ulyanovsk Oblast

IPD SHARING:
Plan to Share IPD: No